CLINICAL TRIAL: NCT02850120
Title: Complications Following Tension-free Vaginal Tape (TVT), Trans-obturator Tape (TOT) and Suprapubic Sling (SS) Procedures for Stress Urinary Incontinence: 8-year Retrospective Cohort Study Using Hospital Episodes Statistics Data
Brief Title: Complications of Mesh Procedures for Stress Urinary Incontinence
Acronym: SUI-mesh
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RX029_MESH_SUI
Record Dates: First submitted 2016-07-18; First posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Urinary Incontinence; Stress
Keywords: surgical mesh; observational study; intraoperative complications; postoperative complications
MeSH Terms: conditions — Urinary Incontinence; Intraoperative Complications; Postoperative Complications | interventions — Suburethral Slings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Unconfounded: All hospital admissions including Tension-free Vaginal Tape (TVT), Trans-obturator tape (TOT) or suprapubic sling (SS) procedures with:
  1. no concomitant procedures,
  2. any concomitant procedures which were considered unlikely to have an effect on outcomes from their mesh insertion, or
  3. only other concomitant procedures which were considered likely to be rescue procedures treating complications caused by the mesh insertion procedure itself.
  Interventions: Procedure: Tension-free vaginal tape (TVT); Procedure: Trans-obturator tape (TOT); Procedure: Suprapubic sling (SS)
- Confounded: All hospital admissions for insertion of Tension-free Vaginal Tape (TVT), Trans-obturator tape (TOT) or suprapubic sling (SS) procedures with concomitant procedures likely to affect outcomes.
  Interventions: Procedure: Tension-free vaginal tape (TVT); Procedure: Trans-obturator tape (TOT); Procedure: Suprapubic sling (SS)

INTERVENTIONS:
Procedure: Tension-free vaginal tape (TVT) — Surgical insertion of Tension-free vaginal tape (TVT) polypropylene mesh in the treatment of stress urinary incontinence.
Procedure: Trans-obturator tape (TOT) — Surgical insertion of Trans-obturator tape (TOT) polypropylene mesh in the treatment of stress urinary incontinence.
Procedure: Suprapubic sling (SS) — Surgical insertion of Suprapubic sling (SS) polypropylene mesh in the treatment of stress urinary incontinence.

SUMMARY:
Complications from mesh procedures (i.e. insertion of tension-free vaginal tapes (TVT), trans-obturator tapes (TOT) and suprapubic slings (SS)) used during surgical treatment of stress urinary incontinence have caused major concern around the world.

The investigators aim to conduct a retrospective cohort study using administrative inpatient data from the Hospital Episode Statistics (HES) database to determine the complications of all first-time surgical mesh procedures in the treatment of stress urinary incontinence (SUI) in women treated in a National Health Service (NHS) hospital in England who were discharged from hospital between 1st April 2007 and 31st March 2015.

The primary outcome measure is the number and types of complications (occurring peri-procedurally, within 30 days of the mesh procedure and those occurring during follow-up). Additional outcomes recorded include: the numbers and types of mesh procedures, including those with potentially confounding concomitant procedures.

ELIGIBILITY:
Inclusion Criteria:

* Women with an Office of Population Censuses and Surveys Classification of Surgical Operations and Procedures 4th revision (OPCS-4) procedure code for an introduction of a Tension-free Vaginal Tape (TVT: M53.3), Trans-Obturator Tape (TOT: M53.6) or Supra-pubic Sling (SS: M52.1) surgical mesh procedure recorded in any of the 24 procedure fields captured in HES, and a recorded diagnosis of stress urinary incontinence based on International Classification of Diseases 10th revision (ICD-10) diagnoses: N39.3, N39.4, R32: T83.1, T83.4, T83.5, T83.6, T83.6, T83.8, T83.9, Z46.6, in any of the 20 diagnosis fields captured in HES.

Exclusion Criteria:

* Duplicate episode of care (exact match on patient identifier; admission date and method; discharge date, destination and method; hospital, gender, age, all procedure codes and all diagnostic codes)
* Male gender
* Missing age
* Aged less than 18 years
* Invalid or missing admission method
* Missing admission date
* Patients with recorded episodes of care in HES which appear after a reported date of death.
* Concomitant mesh surgery for pelvic organ prolapse surgery, or surgical mesh repair, removal, renewal or subsequent mesh insertion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women receiving surgical mesh intervention in the treatment of stress urinary incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 101081 (Actual)
Dates: Start 2007-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Long-term complications | Longitudinal analysis of all episodes of care available in HES (up to 96 months)
  Readmission for further mesh surgery or for symptoms indicating complication

SECONDARY OUTCOMES:
Type of mesh used | Longitudinal analysis of all episodes of care available in HES (up to 96 months)
  Frequency of each type of mesh procedure (TVT, TOT, SS) used over time
Frequency of treatment-related adverse events during initial hospital stay for mesh insertion procedure | During hospital admission when surgical mesh was inserted (length of hospital stay can vary between patients from 0-100 days)
  Frequency of complication
Nature of treatment-related adverse events as determined by clinical coding practice of ICD-10 codes (Aylin et al. BMJ. 2004) | During hospital admission when surgical mesh was inserted (length of hospital stay can vary between patients from 0-100 days)
  Nature of complication
Frequency of 30-day complications | Occurring within 30 days of surgical mesh insertion procedure
  Frequency and nature of complication
Nature of treatment-related adverse events occurring within 30 days of mesh procedure as determined by clinical coding practice of ICD-10 codes (Aylin et al. BMJ. 2004) | Occurring within 30 days of surgical mesh insertion procedure
  Nature of complication

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sims, PhD, Principal Investigator — Newcastle upon Tyne Hospitals NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
Hospital Episode Statistics data to reproduce results are available from the Health and Social Care Information Centre (HSCIC) via formal application process. Analytic code and its output will be shared.